CLINICAL TRIAL: NCT01206374
Title: Demographic and Laboratory Data Collection for Patients With Vitiligo Vulgaris
Brief Title: Questionnaire and Laboratory Data on Vitiligo Vulgaris
Status: Completed | Type: Observational
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-027SLRHC
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Vitiligo Vulgaris
Keywords: Vitiligo Vulgaris
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Vitiligo vulgaris is an autoimmune disorder that causes loss of pigmentation over the skin, hair and mucous membranes (e.g. lips, nose, genitals). While genes have been identified that are thought to be required for development of vitiligo, only 5-10% of relatives develop disease. The triggers for disease onset have not yet been identified. The intent of this study is to research trends in laboratory data, social and medical history that may be contributory to vitiligo onset, location of disease, course of illness and response to therapy.

DETAILED DESCRIPTION:
Patients who participate in this study will be asked to complete a survey and have blood/ laboratory testing performed that relates or may relate to the diagnosis of vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Vitiligo Vulgaris
* Ability to sign consent

Exclusion Criteria:

* Pregnant
* Inability to sign consent
* Inability to complete questionnaire

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients willing to sign consent, complete questionnaire and/ or laboratory studies.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Quality of life disturbances in people with vitiligo | point prevalence
  dermatology life quality indices were you used and correlated with location of disease

SECONDARY OUTCOMES:
self-reporting of vitiligo disease symptoms and history | single survey
  Correlation of the patient survey response with chart documentation was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Nanette Silverberg, MD, Principal Investigator — StLukesNY
Locations (2):
- United States (2):
  - Department of Dermatology, Beth Israel Medical Center, New York, New York
  - Department of Dermatology, St. Luke's-Roosevelt Hospital Center, New York, New York

REFERENCES:
- [Background] Silverberg NB. Update on childhood vitiligo. Curr Opin Pediatr. 2010 Aug;22(4):445-52. doi: 10.1097/MOP.0b013e32833b6ac3. PMID 20616733
- [Background] Silverberg JI, Silverberg AI, Malka E, Silverberg NB. A pilot study assessing the role of 25 hydroxy vitamin D levels in patients with vitiligo vulgaris. J Am Acad Dermatol. 2010 Jun;62(6):937-41. doi: 10.1016/j.jaad.2009.11.024. PMID 20466170
- [Background] Pagovich OE, Silverberg JI, Freilich E, Silverberg NB. Thyroid abnormalities in pediatric patients with vitiligo in New York City. Cutis. 2008 Jun;81(6):463-6. PMID 18666385